CLINICAL TRIAL: NCT02351349
Title: MULTIDISCIPLINARY INTERVENTION FOR FRAIL ELDERLY PATIENTS WITH STAGE 4 or 5 Chronic Kidney Disease (Not on Dialysis)
Brief Title: Chronic Kidney Disease Among Frail Elderly
Acronym: FRED-CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameena Iqbal (Other)
Responsible Party: Sponsor-Investigator, Sameena Iqbal, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-275-GEN
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Chronic Kidney Disease
Keywords: frailty; CKD; Physical Therapy Modalities; Elder Nutritional Physiological Phenomena
MeSH Terms: conditions — Renal Insufficiency, Chronic; Frailty | interventions — Physical Therapy Modalities; Nutrition Therapy; Palliative Care

STUDY DESIGN:
Intervention Model Description: allocated intervention to those who were willing to complete the exercise program due to the difficulty for recruitment, this study was changed to a feasibility study
Oversight: Data Monitoring Committee: No

ARMS (2):
- multidisciplinary intervention (Experimental): Due to the problem of randomization, the study became a before and after assessment in the one group that completed the 12 week exercise program and received nutritional support
  Interventions: Other: multidisciplinary intervention
- Non adherence (No Intervention): Those who were offered the program but did not complete the prescription

INTERVENTIONS:
Other: multidisciplinary intervention — multidisciplinary intervention
  Other Names: physiotherapy; nutritional therapy; supportive therapy
  Arms: multidisciplinary intervention

SUMMARY:
Chronic kidney disease is a common diagnosis in the elderly population and it is associated with significant morbidity and health care costs. The prevalence rates increase with age to about 40% for adults aged > 65 years. In the elderly population (age 65 and over), CKD is associated with a higher burden of comorbid conditions and frailty. The prevalence of frailty is higher in CKD patients with rated being double in early stages and nearly 6 times higher beyond stage 3b. Previously reported frailty mortality rates of 18% at 3 years and 47% at 7 years comparing with mortality rates in non frail individuals of 3% and 12% respectively. In this study, the investigators investigate the effect of multidisciplinary interventions upon frail elderly patients with CKD not yet on dialysis. This interventions include best medical care, nutrition, physiotherapy, and social, psychological and spiritual support.

DETAILED DESCRIPTION:
A multilevel, multidisciplinary intervention is required to assist frail CKD patients given the complexity of their condition. However, the optimal methods for this intervention are not very well defined in the literature.

It was previously described that dialysis does not improve (and often times can worsen) the outcomes of frail patients with renal disease (41). The nowadays trend is to try to optimise and decrease frailty before initiation of dialysis. If that is not possible, a more conservative and palliative approach is envisaged. Regardless, a combined geriatric and nephrological expertise may help to identify patients at high risk of early death for whom this approach is indicated (42).

Major medical societies have regularly reviewed and published their guidelines for medical management of chronic kidney disease. Most reputable such guidelines are KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease (43) and The National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF KDOQI, (44)). In Canada, field experts reviewed current evidence and provided similar recommendations (45). In summary, all this guidelines provide expert opinion on treatment and targets of treatment in CKD patients with an accent on controlling cardiovascular risk factors (hypertension, diabetes, dyslipidemia), lifestyle management, control of CKD complications (proteinuria, anemia, mineral metabolism), and initiation of renal replacement therapy.

Lifestyle management is probably one of the most important intervention in CKD population. First and foremost, it empowers the patients to take control of their lives and become an active partner in their treatment. Smoking cessation, weight reduction, dietary protein control, alcohol intake, exercise, and controlling salt intake are proven to improve outcomes and are part of current guidelines. Regular physical exercise improves physical fitness, walking capacity, cardiovascular parameters (e.g. blood pressure and heart rate), health-related quality of life, and nutritional parameters (48). Physical activity is also protective against depression (49). In the case of frail patients, usually sedentary, with multiple cardiac risk factors, it is recommended to begin with gradual exercise and under supervision.

Nutrition must be targeted in the frail elderly with CKD because decreasing energy intake is associated with higher stages of CKD (50). Though in the CKD non dialysis population, nutrition supplementation has not been formally assessed, the general population of frail elderlies have been evaluated with protein supplementation.

Tieland et al (51) randomized 65 frail elderly in protein versus placebo supplementation groups for 24 weeks. January 11, 2015 revised The protein supplementation group had no benefit with respect to weight gain or muscle strength. However, when resistive exercise training was coupled with protein supplementation, body weight gain was achieved.

Furthermore, Tieland et al (52) randomized 62 frail elderly in two groups, both who received exercise training but only one group received protein supplements. A 0.7 kg weight gain was recorded in the protein supplement but none in the control group. The sustainability and the benefit in survival of such weight gain has not been determined, especially in the CKD non dialysis patients. Thus, the investigators propose that exercise with protein supplementation will benefit the CKD frail older population.

Frail patients with or without CKD are at risk of experiencing psychological distress. Acknowledging one's own limitations, inability to perform up to certain social standards, losing function when comparing with friends or family members within same age group, depending on other's support can all be envisage as high risk factors for depression and/or other psychological ailments. Psychological distress is associated decrease quality of life of worse outcomes. Anxiety and depression are 2 major compounds of psychological distress. Patients can be screened with two easy to use scales: GAD-7 (for anxiety) and PHQ-9 (for depression). Were identified, these conditions should be treated by Psychiatry or Geriatrics services.

Disability is best assessed using the standard ten variables addressed in the Barthel scale (56) are: presence or absence of fecal incontinence, presence or absence of urinary incontinence, help needed with grooming, help needed with toilet use, help needed with feeding, help needed with transfers (e.g. from chair to bed), help needed with walking, help needed with dressing, help needed with climbing stairs, and help needed with bathing. The Maryland State Medical Society holds the copyright for the Barthel Index. It may be used freely for noncommercial purposes with the following citation: Mahoney FI, Barthel D. "Functional evaluation: the Barthel Index." Maryland State Med Journal 1965;14:56-61. The scale is detailed in Appendix 2 and it is used with permission.

Interventions targeted to improve frailty are limited by the patient's ability to collaborate and work with the treating team. Severe cognitive impaired patients lack insight and capacity and they are limited in their capacity to rehabilitated. MoCA (57) is a well validated tool at identifying cognitive impairment, it is widely available in many languages, and it is recommended by The Canadian Consensus Guidelines for Diagnosis and Treatment of Dementia for detection of Mild Cognitive Impairment and Alzheimer's disease. A cut-off of > 17 is generally used to exclude severe dementia. A language specific MoCA and instructions to administer the test are available online at http://www.mocatest.org/. The original English version is reproduced in Appendix 3.

The primary objective of the proposed study is to assess the effect of intensive multidisciplinary interventions on survival, hospitalization and need to start dialysis. Secondary objectives include the assessment of the intervention in different stages of sarcopenia and measurement of physical functioning and nutritional parameters to evaluate the effect of such interventions among the frail CKD population.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must be ≥65 years as of December 2014, with estimated glomerular filtration rate (eGFR) of ≤30ml/min, and experiencing frailty defined as 3 out of 5 criterias: unintentional weight loss (self-reported or January 11, 2015 revised objective 10 lbs in past year)
* Self-reported exhaustion
* Weakness (measured by grip strength)
* Slow walking speed (measured by the 6 minute walking test)
* Low physical activity.

Exclusion Criteria:

* Exclusion criteria are: persons aged <65
* Unable to grasp dynamometer due to various reasons
* Expected life expectancy <6 months due to a non-renal cause
* Patient refusal to participate
* Plan to travel or transfer treatment site during study period and unable to be contacted
* Severe cognitive impairment (as screened with MoCA <18).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameena Iqbal, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill UNiversity Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For recruitment 14 were consented 5 patients dropped out -- 3 started hemodialysis the first week of starting the study and 2 due to medical illness and desire not to follow up with testing
Groups:
- Intervention: Multi Intervention: Due to the problem of randomization, the study became a before and after assessment in the one group that completed the exercise program and received nutritional support
  multidisciplinary intervention: multidisciplinary intervention
- Control: These individuals did not receive exercise advice and did not see the dietician unless there was a clinical problem
Period: Overall Study
Arm/Group | Intervention: Multi Intervention | Control
Started | 6 | 8
Completed | 4 | 5
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Control: Those who were offered the program but did not complete the prescription
- Total: Total of all reporting groups
Arm/Group | Multidisciplinary Intervention | Control | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] — years mean and standard deviation
  years
    Age | 76.5 [69 to 91] | 78 [68 to 85] | 78 [68 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 3 | 5
Weight [Median (Inter-Quartile Range); unit: kilograms] | 67 [60 to 104] | 74 [66 to 102] | 73 [60 to 104]
height [Median (Inter-Quartile Range); unit: meters] | 1.64 [1.52 to 1.79] | 1.63 [1.47 to 1.79] | 1.63 [1.47 to 1.79]
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.2 [21.7 to 32.25] | 29.2 [23.1 to 38.8] | 28.2 [21.7 to 38.8]
estimated GFR [Median (Inter-Quartile Range); unit: ml/min/1.73m^2] | 32 [26 to 39] | 17 [13 to 47] | 31 [13 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: the entire sample will be followed until time of death or until study completed. The cause of
  death will be determined from proxies or from hospital records.
Time Frame: 6 months
Population: mortality
Measure: Number; unit: percentage of mortality
Groups:
- Control: those who were randomized to no exercise program
Arm/Group | Intervention: Multi Intervention | Control
Number analyzed (Participants) | 4 | 5
percentage of mortality | 0 | 0

2. Secondary Outcome: Number of Patients Progressed to the Need for Renal Replacement Therapy (Any Modality or Palliation).
Description: Number of patients progressed to the need for renal replacement therapy (any modality or palliation).
Time Frame: 6 months
Population: three individuals started hemodialysis within 1 week of randomization, they were excluded
Measure: Count of Participants; unit: Participants
Groups:
- Control: those who were not randomized to the exercise group
Arm/Group | Intervention: Multi Intervention | Control
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

3. Secondary Outcome: Hospitalizations
Description: information about principal diagnosis, number and length of hospitalizations will be collected at 6-month intervals from participant, from proxies
Time Frame: 6 months
Population: no hospitalizations recorded in either arm
Measure: Number; unit: participants
Groups:
- Control: those who were not in the exercise group
Arm/Group | Intervention: Multi Intervention | Control
Number analyzed (Participants) | 4 | 5
participants | 0 | 0

4. Secondary Outcome: Physical Functioning Measures
Description: assessed by applying the data of the 4 meter walk compared between the two study groups.
Time Frame: 12 weeks
Population: data on 4m walk, time up and go, dominant hand grip
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Intervention: Multi Intervention | Control
Number analyzed (Participants) | 4 | 5
seconds
  baseline 4 m walk | 5 [3.3 to 7.0] | 5.3 [4.3 to 5.8]
  4m walk at 12 weeks | 3.9 [2.6 to 6.0] | 5.5 [4.2 to 6.2]
Statistical Analysis 1: Comparison: Intervention: Multi Intervention; Test type: Other — paired t test pre compared to post readings; p = 0.0143, t-test, 2 sided

5. Secondary Outcome: Time up and go
Description: one of the physical functioning parameters
Time Frame: 12 weeks
Population: time up and go
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Control: Those who were randomized not to the exercise program
Arm/Group | Multidisciplinary Intervention | Control
Number analyzed (Participants) | 4 | 5
seconds
  baseline | 12 [8.6 to 17.5] | 13 [11.1 to 14.4]
  12 weeks | 10.8 [6.9 to 15.8] | 13.3 [11.3 to 15.5]
Statistical Analysis 1: Comparison: Multidisciplinary Intervention; pre and post comparison of time up and go in intervention group; Test type: Other — as above; p = 0.1416, t-test, 2 sided

6. Secondary Outcome: Dominant Hand Grip
Description: right hand grip average of three values
Time Frame: 12 weeks
Population: paired t test
Measure: Median (Inter-Quartile Range); unit: kg
Groups:
- Control: Those who were randomized not to the exercise group
Arm/Group | Multidisciplinary Intervention | Control
Number analyzed (Participants) | 4 | 5
kg
  baseline | 23 [14 to 35] | 19 [16 to 23]
  12 weeks | 26.5 [14 to 39] | 20 [16 to 28]
Statistical Analysis 1: Comparison: Multidisciplinary Intervention; pre and post value comparison with paired t test was carried out; Test type: Other; p = 0.9013, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The adverse event happened at the time of randomization in the first three months. There was break in randomization technique. The functional outcome testing was only completed at 12 weeks. No testing was done at 24 weeks.
Groups:
- Control: those who were randomized to the no exercise group
Arm/Group | Intervention: Multi Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No